CLINICAL TRIAL: NCT02189356
Title: Evaluation of the Efficacy of an Exercise Program for Pregnant Women With Low Back and Pelvic Pain: A Prospective Randomized Controlled Trial
Brief Title: Gulhane Military Medical Academy Ethical Committee Exercise Program for Pregnant Women With Low Back and Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Ozdemir, PhD, RN, PhD, RN, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1491-348-11/1539-227; GMMA (Other: GMMA)
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Pregnant; Pregnancy-related Low Back and Pelvic Pain
Keywords: Pregnancy-related low back and pelvic pain; exercise program; nurse
MeSH Terms: conditions — Pelvic Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise programme (Experimental): The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Forty-eight pregnant participants with pregnancy-related LBPP were included in the control group and 48 pregnant participants with pregnancy-related LBPP were included in the intervention (exercise) group.
  Interventions: Behavioral: exercise programme
- contol group (Other): The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Forty-eight pregnant participants with pregnancy-related LBPP were included in the control group and 48 pregnant participants with pregnancy-related LBPP were included in the intervention (exercise) group.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: exercise programme — The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Forty-eight pregnant participants with pregnancy-related LBPP were included in the control group and 48 pregnant participants with pregnancy-related LBPP were included in the intervention (exercise) group
  Arms: exercise programme
Behavioral: standard care — standard pregnancy follow up
  Arms: contol group

SUMMARY:
The aim of this study was to evaluate the effect of exercise programs on pregnant women with pregnancy-related Low Back and Pelvic Pain (LBPP). Hypotheses of the study were: 1) Exercise programs relieve the intensity of LBPP in pregnant women and 2) Exercise programs promote functional capacity for pregnant women with LBPP.

DETAILED DESCRIPTION:
Design The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Forty-eight pregnant participants with pregnancy-related LBPP were included in the control group and 48 pregnant participants with pregnancy-related LBPP were included in the intervention (exercise) group.

Participants This research was performed between December 2011 and May 2012 at the Department of Obstetrics and Gynecology, Gulhane Military Medical Education and Research Hospital in Ankara, Turkey. Approximately 3,000 births occur annually at this clinic. Participants were pregnant women who presented to the obstetrics department for routine pregnancy examinations, had pregnancy-related LBPP and fulfilled the eligibility criteria. Eligibility criteria of the research were determined following a literature review. The eligibility criteria were;

* Age over 18 years old
* Ability to read and write in Turkish,
* Volunteering to participate in the study,
* Being between 20-35 weeks of gestation,
* Having no complications for any reason during the study,
* No diagnosis of low back and/or pelvic disease prior to pregnancy,
* Not performing exercise for half an hour at least three days a week during pregnancy,
* Not using analgesics for low back and pelvis pain,
* Not using other methods for the treatment low back and pelvic pain,
* Giving birth before the completion of the study Interventions Participants diagnosed with pregnancy-related LBPP by a doctor and with no medical obstacles to participation in the study were directed to nurse. The nurse invited the pregnant women to the research room for a discussion about low back and pelvic pain. After the eligibility criteria of the pregnant women were reviewed, initial assessments were completed and the participants were subsequently randomized.

The nurse gave health counseling to the participants in the intervention group about the prevention of pregnancy-related LBPP and initiated an exercise program that included exercise training. The health counseling and exercise training booklets provided were prepared based on the literature. Each counseling session lasted an average of 45 minutes. Sessions were completed in a positive education atmosphere and were face-to-face as consistent with the principles of adult education. The structure and function of the vertebrae, physical changes occurring during pregnancy, causes of pregnancy-related LBPP, the problems that the pain causes, methods of pain management, correct posture development, body mechanics during activities of daily life and ergonomics were explained to the pregnant women using illustrated booklets given during the trainings. During the counseling, the nurse received information from the participants regarding their daily activities and educated the participants about the behaviors that might damage the low back and pelvic regions. Participants were given practical demonstrations of how to move and how to protect the low back and pelvic regions during daily life. For example, the nurse demonstrated how to retrieve an object from the ground, how to reach shelves, how to sit and stand up and how to lie down, guiding the participants through these activities as well. The participants' questions were answered, and they were given educational booklets. Following the health consultation, exercise education was given. The participants were given illustrated booklets explaining the effects of pregnancy exercises on maternal and fetal health, situations that need attention before starting and during exercises, signs of danger, what should be done in potentially dangerous situations, how to breathe during exercise and the method, frequency and amount of the exercise. The exercises given to the intervention group were based on the guidelines from "Exercise in Pregnancy" by the Royal College of Obstetricians and Gynaecologists (RCOG) and the guidelines from "Pregnancy and Exercise" by Hacettepe University in Turkey. It was emphasized that pregnant women should complete their exercises as shown at least three days a week for 30 minutes. The duration of the exercise program was four weeks. Participants were offered a choice of two types of exercise according to the weather conditions. The first option comprised exercises performed on a mattress, including stretching, tightening and loosening movements that targeted large muscle groups from the neck to the vertebrae. The nurse explained that the mattress exercises would start with a 5 minute warm up, continue for at least 15-20 minutes at mid-tempo and end with a 5 minute cool down. The second option was a walking exercise. The participants were expected to warm up for 5 minutes, increase their speed for 5 minutes, continue at mid-tempo for 15 minutes and complete a 5 minute cool down. It was emphasized that the pulse rate should be between 120-160/min when the participants reached mid-tempo. In this exercise program, we assumed that both the walking exercise and the mattress exercises had equal effects on the low back and pelvic pain. Pregnant women were able to choose the type of exercise according to their wishes and requirements and could use either or both of the exercise options. The nurse determined the exercise plan with the pregnant women, creating an individual exercise program according to the patient's personal characteristics. The participants were asked to record the type and the duration of the completed exercises during the program on the data collection form and were asked to note if they encountered any problems during the program. The nurse taught the participants how to fill out the forms and answered any questions about the programs. The nurse spoke with the pregnant women on the phone three times a week and gave counseling according to their needs. During interviews, pregnant women were reminded to complete the data collection forms. After four weeks, the researchers made a final assessment of the pregnant women and collected the forms during a face-to-face interview. The exercise programs were terminated at this point, though the pregnant women were able to continue the counseling if they wished.

The pregnant women in the control group received usual care, comprised of routine clinical practice for pregnancy-related LBPP. The control group participants were recommended bed rest and analgesics for LBPP and were not given any treatment for LBPP in addition to standard care. Pregnant women in the control group did not exercise before the study or during the study. The nurse spoke with the women in the control group on the phone once a week and asked them to assess their LBPP and complete the data collection form. The final assessments of the participants were made during a face-to-face interview four weeks later. Willing pregnant women in the control group were advised on pain management strategies after completion of the four weeks of the study.

Sample size and statistical power considerations The sample size was calculated using the PS Software: Power and Sample Size program. Using the literature, we calculated that a sample size of 48 pregnant women in both the exercise group and the control group (total 96 pregnant women) could allow for detection of a difference in VAS score of 10 mm between the intervention and control group, given a SD of 15 mm with accompanying 0.95% confidence intervals (CI) and a power of 0.90.

Randomization According to the CONSORT requirements, the participants were randomly allocated to either the intervention group (n=48) or the control group (n=48) using opaque, sealed envelopes and a simple randomization method. The nurse at the clinic randomly drew the envelopes and broke the seal in the nursing room. The nurse explained the study's purpose and procedures to the pregnant women in the control and intervention groups. The same procedure was repeated for all the pregnant women. Blinding of participants was not feasible due to the study design.

Primary outcomes The primary outcomes of this study were the change in pain intensity at the end of four weeks compared with the baseline and the changes in functional status at the end of weeks first and fourth.

Data collection The nurse collected the data by meeting with the pregnant women at the beginning and end of the study for a total of two interviews. The data collection form included the sociodemographic characteristics of the pregnant women, their pregnancy history, and questions regarding any history of pain. In these meetings the nurse measured the severity of the LBPP and determined the functional status of the pregnant women. The participants measured the severity of LBPP at the end of each week for a total of 4 measurements and recorded their pain on a "Weekly Pain Follow-up Form". Additionally, participants in the intervention group recorded their exercises on a "Daily Exercise Form". The forms were collected for evaluation by the nurse at the completion of the study.

Measures Pain Intensity We used the Visual Analogue Scale (VAS) to measure the intensity of the participants' pain. The VAS is a reliable and valid scale that widely used all over the world for the assessment of pain intensity. Pregnant women noted the severity of the low back and pelvic pain that they perceived on a 100 mm VAS. The nurse determined the intensity of pain by measuring the point the pregnant woman had marked with a ruler. We examined the intensity of two types of pain; perceived pain intensity at rest as VASrelaxation and perceived pain intensity during activity as VASactivity.

Functional Level The Oswestry Disability Index (ODI) was used to determine the participants' functional status. The ODI was developed in 1976 by O'Brien and is a condition-specific outcome measure used in the management of spinal disorders. The ODI has been broadly tested and was found to have good psychometric properties and to be useful in a wide variety of settings. The ODI is the 'gold standard' for low back functional outcome instruments, is self-administered and consists of a 10-item questionnaire. The first section evaluates the intensity of pain and the others describe its disabling effects on typical daily activities including personal care activities (washing, dressing), lifting, walking, sitting, standing, sleeping, social life and travelling. Each item is scored from 0 to 5, with higher values demonstrating greater disability. The ODI's validity and reliability in the Turkish population was examined by Yakut et al. (2004) and the Cronbach α value was reported as 0.91.

Exercise Level Exercise diaries are easy, cost-effective and frequently used methods to measure physical activity. In this study, exercise diaries were used to determine the exercise levels of participants in the intervention group. Exercise for 30 minutes at least 3 days a week was considered sufficient.

Ethical Considerations An Academy Ethical Committee approved the study design, protocols and informed consent procedure with number 1491-348-11/1539-227. Participants were informed about the study before inclusion and could decline to participate at any time. The participants read and signed the informed consent form with the help of the nurse at the beginning of the study.

Data Analysis Based on the intention-to-treat principle, all pregnant women were analyzed according to the group they were assigned to, regardless of whether they received the intervention or not. Missing data were not imputed. To investigate the differences between the groups, the Student's t test was used for values with a normal distribution and the Mann-Whitney U test was used for values without a normal distribution. To investigate the differences within the groups, the paired samples t test was used for values with a normal distribution and the Wilcoxon test was used for values without a normal distribution. Repeated measurement results that did not have a normal distribution were analyzed using the Friedman Test. The error level for all analysis was set at p = 0.05. The results were analyzed using SPSS, version 15.0 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
* Age over 18 years old
* Ability to read and write in Turkish,
* Volunteering to participate in the study,
* Being between 20-35 weeks of gestation,
* Having no complications for any reason during the study,
* No diagnosis of low back and/or pelvic disease prior to pregnancy,
* Not performing exercise for half an hour at least three days a week during pregnancy,
* Not using analgesics for low back and pelvis pain,
* Not using other methods for the treatment low back and pelvic pain,
* Giving birth before the completion of the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pain intensity | 4 weeks
  We used the Visual Analogue Scale (VAS) to measure the intensity of the participants' pain. The VAS is a reliable and valid scale that widely used all over the world for the assessment of pain intensity (Wewers & Lowe 1990, Lindseth & Vari 2005, Kalus et al. 2008, Potter 2013, Murphy et al. 2009).

SECONDARY OUTCOMES:
The Oswestry Disability Index | 4 weeks
  The Oswestry Disability Index (ODI) was used to determine the participants' functional status. The ODI was developed in 1976 by O'Brien (Fairbank & Pynsent 2000) and is a condition-specific outcome measure used in the management of spinal disorders.

REFERENCES:
- [Derived] Ozdemir S, Bebis H, Ortabag T, Acikel C. Evaluation of the efficacy of an exercise program for pregnant women with low back and pelvic pain: a prospective randomized controlled trial. J Adv Nurs. 2015 Aug;71(8):1926-39. doi: 10.1111/jan.12659. Epub 2015 Mar 31. PMID 25823561